CLINICAL TRIAL: NCT05334823
Title: A Phase II Clinical Study of Anti-CD19 CAR-T Therapy (pCAR-19B) in the Treatment of CD19-positive Relapsed/Refractory B-ALL
Brief Title: A Study of pCAR-19B in the Treatment of CD19-positive Relapsed/Refractory B-ALL in Children and Adolescents
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PB07
Record Dates: First submitted 2022-03-16; First posted 2022-04-19 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Acute Lymphoblastic Leukemia; Relapsed Pediatric ALL; Refractory Acute Lymphoblastic Leukemia
Keywords: CAR-T; CD19; B-ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pCAR-19B cells (Experimental): Infusion of pCAR-19B cells by dose of 0.6-2 x106 cells/kg
  Interventions: Biological: pCAR-19B cells

INTERVENTIONS:
Biological: pCAR-19B cells — Drug: pCAR-19B cells； Administration method: intravenous infusion； Subjects will be treated with Fludarabine and Cyclophosphamide before cell infusion.

SUMMARY:
This is a phase II clinical study to evaluate the safety and efficacy of pCAR-19 B cell autologous infusion preparation in the treatment of CD19-positive relapsed/refractory B-cell acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
This is a multiple-center, single-arm, open-label study. After meeting the eligibility criteria and enrolling on the trial, patients will undergo leukapheresis for collection of autologous lymphocytes. Once cells have been manufactured, patients will then proceed to lymphodepleting chemotherapy with cyclophosphamide 300mg/m2 and fludarabine 30mg/m2 for 3 consecutive days followed by the infusion of CD19 CAR T-cells at a target dose of 0.6-2 x106 cells/kg.

ELIGIBILITY:
Inclusion Criteria:

1. The patient himself or his guardian agrees to participate in this clinical trial and signs the Informed Consent Form (ICF), indicating that he understands the purpose and procedures of this clinical trial and is willing to participate in the research;
2. Diagnosed with B-ALL，and meet one of the following conditions:

   1. Refractory B-ALL: early-stage refractory patients who failed to achieve complete remission after 2 courses of standard induction chemotherapy;
   2. Relapsed B-ALL: patients with early relapse (<12 months) after complete remission;or late relapse (≥12 months) after complete remission, and relapsed patients who have not achieved complete remission after standard treatment or have poor response to early treatment; experience Patients with 2 or more bone marrow recurrences; patients with recurrence after allogeneic hematopoietic stem cell transplantation;
   3. For Ph+ALL patients, patients who have not achieved complete remission after receiving at least two Tyrosine kinase inhibitors (TKI) treatments or have relapsed after complete remission (except those who cannot tolerate TKI treatment or have contraindications to TKI treatment or have T315i mutation resistance to TKI drugs);
3. The malignant cells in the bone marrow were confirmed to express CD19 by flow cytometry;
4. Bone marrow morphology at the time of screening indicated that blasts≥ 5%;
5. Eastern Cooperative Oncology Group (ECOG) 0-1 points ;
6. Expected survival is ≥ 12 weeks;
7. The function of important organs is basically normal:

   1. Cardiac function: echocardiography showed cardiac ejection fraction ≥50%, and no obvious abnormality was found on electrocardiogram;
   2. Renal function: serum creatinine≤2.0×ULN;
   3. Liver function: Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤5.0×ULN;
   4. Total bilirubin≤2.0×ULN (for Gilbert syndrome, total bilirubin≤3.0×ULN);
   5. Blood oxygen saturation≥92% in non-oxygen state.
8. No serious mental disorder;
9. Have apheresis or venous blood collection standards, and have no other contraindications for cell collection;
10. Subjects of childbearing age agree to use reliable and effective contraceptive methods for contraception (excluding rhythm contraception) from signing the informed consent to receiving pCAR-19B cell infusion within 1 year.

Exclusion Criteria:

1. Relapse of isolated extramedullary disease;
2. Active central nervous system leukemia at screening, defined as Central Nervous System (CNS)-grade 2 and 3 according to National Comprehensive Cancer Network (NCCN) guidelines (note: those with central nervous system involvement but improved after treatment can be included);
3. Those who have received CAR-T therapy or other gene-modified cell therapy before screening;
4. Received anti-CD19 drug treatment before screening;
5. Received the following anti-tumor treatments before screening: Received chemotherapy, targeted therapy and other drug treatments within 14 days or at least 5 half-lives (whichever is shorter); Received radiotherapy within 14 days;
6. HBsAg or HBcAb positive and hepatitis B virus (HBV) DNA is greater than the normal range; hepatitis C virus (HCV) antibody is positive and HCV RNA greater than the normal range; HIV antibody positive; syphilis positive; Cytomegalovirus (CMV) DNA positive;
7. Have any of the following heart conditions:

   1. New York Heart Association (NYHA) stage III or IV congestive heart failure;
   2. Myocardial infarction or coronary artery bypass grafting within 6 months prior to enrollment (CABG);
   3. Clinically significant ventricular arrhythmia, or history of syncope of unknown origin (by vasovagal except those caused by menstruation or dehydration);
   4. History of severe non-ischemic cardiomyopathy;
8. Active infection or uncontrollable infection requiring systemic treatment within 1 week before screening;
9. The presence of grade 2-4 acute graft-versus-host disease (GVHD) or moderate to severe chronic GVHD within 4 weeks before screening;
10. Cerebrovascular accident or epileptic seizure within 6 months before screening;
11. Active autoimmune diseases；
12. Patients with malignant tumors other than acute lymphoblastic leukemia within 5 years before screening, except for fully treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical resection, and duct in situ after radical resection cancer;
13. Received live attenuated vaccine within 4 weeks before screening;
14. Participated in other interventional clinical studies before screening, including: the last use of unmarketed new drugs is less than 3 months from the time of cell reinfusion, or the last use of marketed drugs is less than 5 half-lives from the time of cell reinfusion;
15. Women who are pregnant or breastfeeding, and male or female subjects who plan to have children within 1 year after receiving pCAR-19B cell reinfusion;
16. Other investigators deem it inappropriate to participate in the study.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-26 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate after pCAR-19B infusion [Effectiveness] | 3 months
  Objective response rate includes CR, CRi.

SECONDARY OUTCOMES:
Minimal residual disease（MRD） | 3 months
  MRD-negative ORR within 3 months by flow cytometry as assessed by Independent Review Committee (IRC) and investigator.
Best overall response after pCAR-19B infusion [Effectiveness] | 2 years
  Best overall response means the proportion of patients with the best efficacy (CR or CRi) after pCAR-19B cell therapy.
Overall survival after pCAR-19B infusion [Effectiveness] | 2 years
  Overall survival means the time from infusion of pCAR-19B cells to death of subjects from any cause
Duration of response after pCAR-19B infusion [Effectiveness] | 2 years
  Duration of response means the time from first assessment of CR or CRi to first assessment of disease recurrence or death from any cause, whichever occurs first
Relapse free survival after pCAR-19B infusion [Effectiveness] | 2 years
  Relapse free survival means time from subject infusion of pCAR-19B cells to first disease relapse or death from any cause (whichever occurs first)
Event free survival after pCAR-19B infusion [Effectiveness] | 2 years
  Event free survival means the time from the infusion of pCAR-19B cells to the time of the following events (whichever occurs first):
  1. Death from any cause after remission;
  2. Disease recurrence;
  3. Withdrawal from the clinical trial after treatment failure or meeting the withdrawal criteria.
The incidence of Treatment Emergent Adverse Events (TEAE) of pCAR-19B infusion | 2 years
  Number of participants with adverse events as assessed by CTCAE v5.0
the incidence of adverse events related to treatment of pCAR-19B infusion | 2 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
the incidence of adverse event of special interest (AESI) of pCAR-19B infusion | 2 years
  Number of participants with special interest adverse events as assessed by CTCAE v5.0,The following adverse events were defined as adverse events of special interest for this study:
  1. Cytokine release syndrome (CRS) of grade 3 and above;
  2. Immune effector cell-associated neurotoxicity syndrome (ICANS) of grade 3 and above;
  3. Grade 3 and above infection;
  4. Grade 3 and above acute tumor lysis syndrome;
  5. Unresolved cytopenias lasting 28 days.
the incidence of RCL of pCAR-19B infusion | 2 years
  RCL Detection: the incidence of Replication Competent Lentivirus.
Pharmacokinetic data parameters of Cmax | 3 months
  Analysis using CAR DNA copy number measured by qPCR: the highest concentration of pCAR-19B cells expanded in peripheral blood after administration
Pharmacokinetic data parameters of Tmax | 3 months
  Analysis using CAR DNA copy number measured by qPCR: the time to reach the highest concentration;
Pharmacokinetic data parameters of AUC0-90d | 3 months
  Analysis using CAR DNA copy number measured by qPCR: Area under the curve at 28 days and 90 days.
Pharmacodynamics data parameters of the degree of clearance | 3 months
  The degree of clearance of CD19-positive B cells at different blood collection time points after cell infusion
Pharmacodynamics data parameters of CAR-T-related serum cytokines | 3 months
  the concentration levels of IL-6 at each time point.
Immunogenicity of pCAR-19B cells | 3 months
  Analysis using anti-CAR antibodies measured by Meso Scale Discovery（Electrochemiluminescence）

OTHER OUTCOMES:
Comparative analysis of 6-month ORR of CAR-T treatment with or without hematopoietic stem cell transplantation | 6 months
  Independent Review Committee (IRC) and investigator-assessed 6-month ORR, including CR and CRi; Independent Review Committee (IRC) and investigator-assessed 6-month ORR with MRD-negative, including CR and CRi.
Assess the Children's growth and development after pCAR-19B infusion | 2 years
  The subject's height were measured before infusion and 1, 2, 3 months after infusion and every three months thereafter.
Assess the Children's growth and development after pCAR-19B infusion | 2 years
  The subject's weight were measured before infusion and 1, 2, 3 months after infusion and every three months thereafter.
The impact of the cellular and molecular features of immune function statu on response and adverse reactions | 3 months
  The correlation between the detection results of peripheral blood lymphocyte subsets which measured by Cellular immunoassay and the efficacy and safety.
Comparative analysis of 6-month RFS of CAR-T treatment with or without hematopoietic stem cell transplantation | 6 months
  6-month relapse-free survival (RFS) by Independent Review Committee (IRC) and investigator assessments was statistically compared between the two groups; Relapse free survival means time from subject infusion of pCAR-19B cells to first disease relapse or death from any cause (whichever occurs first).
Comparative analysis of 6-month OS of CAR-T treatment with or without hematopoietic stem cell transplantation | 6 months
  6-month Overall survival (OS) by Independent Review Committee (IRC) and investigator assessments was statistically compared between the two groups; Overall survival means the time from infusion of pCAR-19B cells to death of subjects from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Tianyou Wang, M.D. Ph.D, Principal Investigator — Beijing Children's Hospital; Yicheng Zhang, M.D. Ph.D, Principal Investigator — Tongji Hospital, Affiliated to Tongji Medical College of Huazhong University of Science and Technology
Locations (10):
- China (10):
  - Beijing Children's Hospital.Capital Medical University, Beijing, Beijing Municipality
  - Beijing GoBroad Boren Hospital, Beijing, Beijing Municipality
  - Pediatric Hematology department of Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiehe Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Xiangya Hospital, Central South University, Changsha, Hunan
  - Children's Hospital Of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - West China Second University Hospital,Sichuan University, Chengdu, Sichuan
  - Institute Of Hematology&Blood Diseases Hospital,Chinese Academy Of Medicai Sciences, Tianjin, Tianjin Municipality